CLINICAL TRIAL: NCT03524885
Title: Standard Implants With Bone Regeneration vs Short Implants (Implantes Convencionales Con regeneración ósea vs. Implantes Cortos)
Brief Title: Standard Implants With Bone Regeneration vs Short Implants
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, David Peñarrocha Oltra, Assistanat Postdoctoral Lecturer (Profesor Ayudante Doctor), University of Valencia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: H1506438508468
Record Dates: First submitted 2018-03-03; First posted 2018-05-15 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Implant Complication; Bone Resorption
MeSH Terms: conditions — Bone Resorption | interventions — Bone Regeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Short implants (Active Comparator): 2 or 3 implant 4-5 mm length and 4 mm diameter (Syra Short, Sweden & Martina, Padua, Italy) will be positioned. The healing cap will be immediately connected and a vycril suture will be done after soft tissue reflection.
  Interventions: Procedure: Short implant placement
- Bone regeneration with longer implants (Experimental): A horizontal and vertical regeneration following GBR technique will be performed using not-resorbable PTFE titanium reinforced membrane (Cytoplast Osteogenics, US) fixed by titanium pins or miniscrews to ensure the perfect stability (Pro-fix, Cytoplast Osteogenics, US).
  The graft will be composed half autogenous bone harvested with a scraper (Meta, Firenze, Italy) by the same surgical site or by a second tunnel site in the mandibular ramus and half deproteinized bovine bone (Bio Oss Geislicht Pharma, Switzerland). The mucosal flaps will be sutured in a double layer with horizontal mattress and single gore-tex sutures (Cytoplast PTFE sutures 3.0, Cytoplast Osteogenics, US).
  2 or 3 implant from 10 to 13 mm length putting the implant platform 2 or 3 mm apical to CEJ of the adjacent tooth will be inserted.
  Interventions: Procedure: Bone regeneration with longer implants

INTERVENTIONS:
Procedure: Short implant placement — Ten patients will be randomly selected for the short implants option, 2 or 3 implant 4-5 mm length and 4 mm diameter (Syra Short, Sweden & Martina, Padua, Italy) will be positioned. The healing cap will be immediately connected and a vycril suture will be done after soft tissue reflection.
  After three months an acrylic screw-retained bridge will be delivered. After further three months, a definitive restauration with a metal ceramic bridge will be seated.
  Arms: Short implants
Procedure: Bone regeneration with longer implants — Ten patients will be randomly assigned to the regenerative group, 2 or 3 implant from 10 to 13 mm length intentionally exposed putting the implant platform 2 or 3 mm apical to CEJ of the adjacent tooth will be inserted.
  A horizontal and vertical regeneration following GBR technique will be performed using not-resorbable PTFE titanium reinforced membrane (Cytoplast Osteogenics, US) fixed by titanium pins or miniscrews to ensure the perfect stability (Pro-fix, Cytoplast Osteogenics, US).
  Arms: Bone regeneration with longer implants

SUMMARY:
A study designed as a randomized controlled trial of parallel group design will be conducted at the Dental clinic of the University of Valencia to compare, considering different parameters, the rehabilitation with dental implants of atrophic posterior mandibles or maxillae using short implants or longer implants with vertical bone regeneration with GBR.

The hypothesis of the study is that both treatment options will be successful to rehabilitate atrophic posterior mandibles or maxillae. Moreover, more surgical complications will be encountered in the bone regeneration group.

ELIGIBILITY:
Inclusion Criteria:

* All the patients with a distal edentulism Kennedy -Applegate Class II in the posterior mandible or maxilla, with residual bone height from the top of the crest to the opposite landmark (the alveolar nerve for the lower and the sinus cavity for the upper) between 5 and 7 millimeters. The bone peak on the last tooth before the edentulous space must be positioned from 2 to 4 mm from the CEJ. (X-ray evaluation by periapical film on a Rinn Holder).
* All patients with at least 3 mm of keratinized tissue on the edentulous crest. In case of absence of this prerequisite, three months before the keratinized tissue is augmented by a ephytelium-connective tissue graft harvested from the palate.
* Patients with edentulous distal sites

Exclusion Criteria:

* Heavy smokers (more than 10 cigarettes /day)
* Patients with active periodontal disease: full mouth plaque index (FMPI > 20%) and Full mouth bleeding index (FMBI > 20%).
* Patients with less of 5 mm of bone width.
* Patients with systemic conditions or under prescription of medications that contraindicate oral surgery

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2018-01-08 (Actual); Primary Completion 2019-07 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Peri-implant bone level changes | 12 months after implant loading
  Interproximal bone level measured on a periapical film taken with a Rinn Holder

SECONDARY OUTCOMES:
Patient satisfaction | 12 months after implant loading
  by means a Visual Analogue Scale ranging between 0 (lowest) and 10 (highest)
Implant survival rate | 12 months after implant loading
  % of implants in function

CONTACTS AND LOCATIONS:
Locations (1):
- Clínica Odontológica de la Universitat de Valencia, Fundación Lluis Alcanyis, Valencia, Spain